CLINICAL TRIAL: NCT05532696
Title: A Phase Ib/II, Open-Label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ABT-101 in Patients With Advanced Solid Tumors and HER2 Exon 20 Insertions Mutated Non- Small Cell Lung Cancer
Brief Title: Phase 1b/2 Study to Evaluate ABT-101 in Solid Tumor and NSCLC Patients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anbogen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT101-102
Record Dates: First submitted 2022-08-30; First posted 2022-09-08 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor; Non Small Cell Lung Cancer; HER2 Mutations
Keywords: ABT-101; NSCLC; HER2 Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABT-101 (Experimental): Part 1- dose-escalation: ABT-101 in patients with advanced cancer disease
  Part 2- dose expansion: ABT-101 in patients with NSCLC with confirmed HER2 mutations
  Interventions: Drug: ABT-101

INTERVENTIONS:
Drug: ABT-101 — Patients will receive ABT-101 by oral administration on a 28-day cycle
  Other Names: DBPR112

SUMMARY:
A Phase 1b/2, open-label, multicenter study to determine the recommended phase 2 (RP2D) of ABT-101in solid tumor and to explore antitumor activities of ABT-101 in patients with HER 2 mutated non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This study will be conducted in two parts:

Part 1: Dose- Escalation, Phase 1b, is designed to determine the RP2D. Patients with solid tumor will be enrolled into a dose finding study scheme with the assessment of dose-limiting toxicities (DLTs). DLT assessment will be conducted during treatment cycle 1

Part 2: Dose- Expansion, Phase 2, will evaluate the safety and efficacy of ABT-101 at the dosage and dosing regime determined in Phase 1b. Phase 2 will enroll NSCLC patients with HER2 mutations

Study participation for all patients includes screening period, treatment period and safety/ follow-up period. Patient will received study treatment until progressive disease or any other discontinuation or withdrawal criterion is met

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 20 years or adult age as per local regulations, at time of informed consent
* Histologically or cytologically confirmed advanced solid tumor (Part 1) or NSCLC with HER2 mutations as determined by the central result (Part 2)
* For patients in Part 2 only: Patients has measurable disease per RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Part 1), 0 to 2 (Part 2)
* Appropriate candidate for experimental therapy
* Adequate organ function

Exclusion Criteria:

* Known active or untreated central nervous system (CNS) metastases and/or carcinomatous meningitis
* For patients in Part 2 only: Previously treated with EGFR or HER2 TKIs.
* Serious acute or chronic infections
* Received a live-virus vaccination
* Received prior anticancer or other investigational therapy within 28 days or 5× the half-life prior to the first dose.
* Not recovered from prior- treatment toxicities to Grade ≤1
* Major surgery within 28 days prior to the study treatment
* Concurrent malignancy within 2 years prior to first dose
* History or presence of clinically relevant cardiovascular abnormalities. QTcF ≥ 470 ms
* Significant gastrointestinal disorder(s) that could interfere with absorption of ABT101
* Known to have a history of alcoholism or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended Phase 2 Dose (RP2D) of ABT-101 in Part 1 | 18 months
  Determine the maximum tolerated dose (MTD) and RP2D of ABT-101 based on Dose Limiting Toxicities
Determine antitumor activity based on Objective Response Rate (ORR) in Part 2 in patients with NSCLC with targeted mutation | 36 months
  Patients response according to RECIST 1.1

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) ABT-101 | 48 months
  Plasma concentration of ABT-101
Area under the plasma concentration time curve (AUC) of ABT-101 | 48 months
  Measure of AUC
Duration of response (DOR) | 48 months
  DOR is defined as the length of time between first response and the date of objectively documented progression of disease or death
Progression- free survival (PFS) | 36 months
  Measure of the time from study entry to disease progression or death due to any cause
Overall survival (OS) | 36 months
  Measure of overall survival
Objective response rate (ORR) in Part 1 | 12 months
  Objective response rate as determined by RECIST 1.1
Disease control rate (DCR) | 36 months
  DCR is defined as the percentage of patients who have achieved a CR, PR, or SD.

CONTACTS AND LOCATIONS:
Locations (5):
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Medical Univresity Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District